CLINICAL TRIAL: NCT07219407
Title: An Open-label, Long-term Study Evaluating RAP-219 in Adult Participants With Refractory Onset Seizures
Brief Title: A Long-term Study of the Safety and Effectiveness of RAP-219 in Adults With Focal Onset Seizures
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rapport Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAP-219-FOS-901
Record Dates: First submitted 2025-10-08; First posted 2025-10-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Focal Epilepsy; Epilepsy; Refractory Focal Epilepsy; Seizure; Focal Seizure; Focal Onset Seizure
Keywords: Focal Seizures; Epilepsy; RNS; Long episode
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Seizures

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RAP-219 (Experimental)
  Interventions: Drug: RAP-219

INTERVENTIONS:
Drug: RAP-219 — Participants will receive one RAP-219 0.125 mg capsule daily for 3 days followed by one 0.25mg tablet RAP-219 daily for 28 days, then one 0.75mg tablet daily for the remainder of the treatment period.

SUMMARY:
This is a clinical research study for an investigational drug called RAP-219 in patients with Refractory Focal Epilepsy. This study is being conducted to determine RAP-219 Long- term safety and open-label antiseizure activity in patients with Refractory Focal Epilepsy.

DETAILED DESCRIPTION:
This is a multi-center, open-label study to evaluate the long-term safety, tolerability, pharmacokinetics, pharmacodynamics and antiseizure activity of RAP-219 in adult participants with refractory focal seizures

ELIGIBILITY:
Inclusion Criteria:

* Completion of the associated parent study (RAP-219-FOS-201) treatment period with acceptable tolerability, per Investigator.
* Diagnosis of refractory focal epilepsy
* Stable RNS(c) system settings
* A demonstrated history of compliance with RNS(c) system data interrogation and upload
* Good overall health other than focal epilepsy, per Investigator.
* BMI ≥ 18 kg/m^2 and ≤ 45 kg/m^2
* Willing and able to adhere to all aspects of the protocol.

Exclusion Criteria:

* Known of hypersensitivity to RAP-219
* Any clinically unstable or serious medical, neurological (other than epilepsy), psychological, or behavioral problem; laboratory or ECG finding that would increase participant risk or should otherwise exclude the patient from participation, as assessed by Investigator
* Pregnancy, lactation, or individuals of reproductive potential who do not agree to simultaneously use two effective birth-control methods

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-02-03 (Estimated); Study Completion 2028-02-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From the start of RAP-219 treatment through 8 weeks after last dose, up to Week 112

SECONDARY OUTCOMES:
Percent change in clinical seizure frequency | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Group median percent change in clinical seizure frequency per 28-day period as reported in a clinical seizure diary
Clinical seizure 25%, 50%, 75%, and 100% responder proportions | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Proportion of participants with at least 25%, 50%, 75%, or with 100% reduction in clinical seizure frequency per 28-day period as reported in a clinical seizure diary
Change in clinical seizure-free day frequency | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Group median change in clinical seizure-free day frequency per 28-day period as reported in a clinical seizure diary
Longest clinical seizure-free interval | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Duration, in days, of the longest continuous period of clinical seizure-free days per period as reported in a clinical seizure diary
Time to pre-randomization clinical seizure count | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Duration, in days, between the beginning of the open-label treatment period and the nth clinical seizure, where n is the number of clinical seizures per 28-day period during the prospective pre-treatment baseline period, as reported in a clinical seizure diary
RNS long episode 30%, 50%, 75% or with 100% responder proportions | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Proportion of participants with at least 30%, 50%, 75%, and 100% reduction in long episodes per 28-day period as recorded by the RNS® System
Percent change in RNS long episode frequency | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Group median percent change in long episode frequency per 28-day period as recorded by the RNS® System
Change in RNS long episode-free day frequency | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Group median change in long episode-free day frequency per 28-day period as recorded by the RNS® System
Longest RNS long episode-free interval | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Duration, in days, of the longest continuous period of long episode-free days per period as recorded by the RNS® System
Time to pre-randomization long episode count | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Duration, in days, between the beginning of the open-label treatment period and the mth long episode, where m is the number of long episodes per 28-day period during the pre-treatment baseline period, as recorded by the RNS® System
Percent change in RNS estimated electrographic seizure frequency | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Group median percent change in estimated electrographic seizure frequency per 28-day period as recorded by the RNS® System
Clinical Global Impression of Change (CGI-C) responder count and proportions | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Count and proportion of participants with any improvement (minimally improved, much improved, or very much improved) or clinically meaningful improvement (much improved or very much improved) as reported on the Clinical Global Impression of Change (CGI-C) scale
Patient Global Impression of Change [PGI-C] responder count and proportions | Throughout the open-label period until 8 weeks after the last dose, up to Week 112, compared to the pre-treatment baseline period.
  Count and proportion of participants with any improvement (minimally improved, much improved, or very much improved) or clinically meaningful improvement (much improved or very much improved) as reported on the Patient Global Impression of Change (PGI-C) scale

CONTACTS AND LOCATIONS:
Overall Officials: Imran Quraishi, MD, Principal Investigator — Yale University
Locations (7):
- United States (7):
  - Consultants in Epilepsy and Neurology, PLLC, Boise, Idaho
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Comprehensive Epilepsy Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania - Department of Neurology, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas